CLINICAL TRIAL: NCT02634450
Title: Evaluation of Point-Of-Care Testing Assays for Early Infant in Mozambique-Cluster Randomised Trial
Brief Title: Early Infant Diagnosis Point of Care Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Saúde, Mozambique (Other Government)
Collaborators: Clinton Health Access Initiative Inc. (Other); UNICEF (Other); UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: POC EID PILOT
Record Dates: First submitted 2015-12-05; First posted 2015-12-18 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: HIV
Keywords: HIV; Diagnostic; children
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Current practice of Early Infant Diagnosis in Mozambique: using conventional system of collecting blood on Dried Blood Spot and sending it to central laboratory for PCR processing and receiving result by SMS printer.
- Intervention (Active Comparator): Point Of Care Device (Alere q) is used for Early Infant Diagnosis, with the sample collected and processed in the consultation room with the device
  Interventions: Device: Alere q

INTERVENTIONS:
Device: Alere q
  Arms: Intervention

SUMMARY:
In Mozambique, early infant HIV diagnosis (EID, i.e. HIV screening of infants under 18 months of age) is conducted using molecular diagnostics at central laboratories in Maputo, Nampula, Beira and Quelimane. However, test volumes are growing and many parts of the country do not have close access to laboratories. Test samples are transported over large distances and this can introduce testing delays, especially for patients in rural and remote areas of the country. There are now new POC EID technologies becoming available that will enable diagnosis of HIV in infants within minutes or a couple of hours on site in the clinic, operated by non technical staff and without laboratory infrastructure. This protocol describes a plan to conduct an evaluation of a Point-Of-Care (POC) Early Infant Diagnosis (EID) testing technologies that are being considered for use in Mozambique, and to pilot those technologies in order to provide more effective diagnostics and clinical care to patients. During this implementation pilot, sites are randomized to use either conventional or POC EID testing only before the inclusion of the patients in the study. No consent will be asked to the parents or guardians. A written permission will be asked to the Direção Provincial de Saúde of both provinces to implement the POC device as routine in those intervention sites. All the information that will be analyzed will be collected from the routine care and it will be analyzed as a group.

ELIGIBILITY:
Inclusion Criteria:

* Born to HIV positive mother
* From 4 weeks to 18 months of age
* Came to CCR consultation for Early Infant Diagnosis

Exclusion Criteria:

* With a valid positive test by other center

Ages: 4 Weeks to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 179 (Actual)
Dates: Start 2015-09; Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
The proportion of HIV-positive infants initiating antiretroviral therapy within 60 days of sample collection | up to 6 months
the proportion of HIV-positive infants who initiated antiretroviral therapy that were retained in care at 90 days of follow-up. | 3 months after treatment initiation
  Patients were considered retained in care at 90 days if they had visited the health facility within the previous 30 days.

SECONDARY OUTCOMES:
The median age at time of results received by patient | Up to 6 months
The median number of days between specimen collection and results received by patient | Up to 6 months
The median age at time of antiretroviral treatment initiation | Up to 6 months
The median number of days between specimen collection and initiation of antiretroviral treatment. | Up to 6 months

CONTACTS AND LOCATIONS:
Locations (8):
- Mozambique (8):
  - Centro de Saude Moamba, Moamba, Maputo Province
  - Centro de Saude de Manga Loforte, Beira, Sofala
  - Centro de Saude de Ponta Gea, Beira, Sofala
  - Centro de Saude Munhava, Beira, Sofala
  - Centro de Saude NHACONJO, Beira, Sofala
  - Centro de Saude de Machava II, Maputo
  - Centro de Saude Matola Gare, Maputo
  - Centro de Saúde de Khongolote, Maputo

REFERENCES:
- [Derived] Jani IV, Meggi B, Loquiha O, Tobaiwa O, Mudenyanga C, Zitha A, Mutsaka D, Mabunda N, Vubil A, Bollinger T, Vojnov L, Peter TF. Effect of point-of-care early infant diagnosis on antiretroviral therapy initiation and retention of patients. AIDS. 2018 Jul 17;32(11):1453-1463. doi: 10.1097/QAD.0000000000001846. PMID 29746301